CLINICAL TRIAL: NCT04406480
Title: Contribution of the Exome Sequencing in Antenatal Period Behind Ultrasound Features Suggestive of a Rare Genetic Disease
Brief Title: Realization of Sequencing of All Known Human Genes in Case of Detection of Cerebral, Renal or Ophthalmological Fetal Malformations During Pregnancy in Order to Make an Etiological Diagnosis and to Precise the Fetal Prognosis
Acronym: PRENATEX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 7344
Record Dates: First submitted 2020-05-26; First posted 2020-05-28 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Fetal Malformation; Pregnancy Related; Rare Genetic Disease
Keywords: Fetal malformations; Exome sequencing; antenatal cerebral malformations; antenatal ocular malformations; antenatal large hyperechoic kidneys
MeSH Terms: conditions — Congenital Abnormalities | interventions — Exome Sequencing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 90 trios (270 subjects: 90 fetus, 90 mothers, 90 fathers) (Other)
  Interventions: Genetic: CGH-array and exome sequencing

INTERVENTIONS:
Genetic: CGH-array and exome sequencing — A blood sample will be used for CGH-array and exome sequencing

SUMMARY:
Congenital malformations concern 3% of pregnancies; most of them can be seen during pregnancy. For some malformations, an invasive sample (trophoblast biopsy or amniocentesis) is proposed to search a chromosomal abnormality by the technique of DNA chip. However, some strongly suggestive signs of a genetic (and not chromosomal) pathology have a very low diagnostic rate with this technique. In the absence of an etiological diagnosis, the prognosis for the unborn child is very difficult to assess, as we can't know if the fetal malformation is really isolated or associted to other unseen features as part of a syndromic condition.

For some malformations strongly suggestive of a genetic condition, we propose to realize an exome (i.e. all coding parts of the genome) sequencing of the trio (child and the 2 parents) with a delivery time compatible with the emergency situation of a pregnancy (6 weeks maximum). We will apply bioinformatics filters to analyse only genes known to be involved in the malformation present in the unborn child and thus avoid the identification of variants in unrelated genes. These lists of genes have been previously validated by the Rare Disease Health Sectors and the affiliated diagnostic laboratories. The selected malformations are: 1) anomalies of the central nervous system (microcephaly (<- 2DS) with anomalies of gyration, anomalies of the posterior fossa, anomalies of the midline except agenesis of the corpus callosum), 2) ophthalmological anomalies (microphthalmia, hyperplasia vitreous) and 3) renal abnormalities (large hyperechoic kidneys).

ELIGIBILITY:
Inclusion Criteria:

* Father and mother of an unborn child past the age of majority
* Consent dated and signed by the mother and by the father
* Father and mother able to understand the objectives and risks of the study
* For the mother, pregnancy in progress (between 12 and 34 weeks)
* For the mother, pregnancy with the presence of a malformation on ultrasound, confirmed by a doctor from the multidisciplinary diagnostic prenatal center, entering into the indications retained for this study
* Clinical validation of the couple's eligibility by an expert for some of selected indications
* Father and mother affiliated to a social protection health

Exclusion Criteria:

* Identified genetic or chromosomal abnormality explaining the observed malformation
* Inability to give informations to the father and / or mother (father or mother in emergency or life-threatening situation)
* Father and / or mother under the protection of justice
* Father and / or mother under guardianship or curatorship
* Nursing woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-08-05 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Diagnostic contribution of the exome sequencing in antenatal period in comparison with the chromosomal analysis (CGH-array) realized in current health care | 13 months
  Comparison of the number of genetic diagnoses made by exome sequencing and by CGH-array.

SECONDARY OUTCOMES:
Effects on pregnancy management and/or postnatal child care due to an etiological diagnosis | 13 months
  Percentage of antenatal and/or postnatal fetus/child care modified by the molecular result
Feasibility study of carrying out exome sequencing in the antenatal period in terms of time to deliver results | 13 months
  Time to results from the inclusion of the trio (in days) specifying the time for each step (reception, sequencing, bioinformatics analysis, interpretation) (in days)

OTHER OUTCOMES:
Difficulties of interpretation of the exome sequencing in antenatal period | 13 months
  Numbers of variants of unknown signification identified by exome sequencing with and without bioinformatic filters (targeted exome)
Identification of new genes responsible of fetal malformations | 13 months
  If the results of CGH-array and targeted exome sequencing are negative, analysis of the entire exome sequencing to find new genes implicated in fetal development

CONTACTS AND LOCATIONS:
Locations (12):
- France (12):
  - CHu de Besançon, Besançon
  - CHU de Dijon, Dijon
  - Hospices Civils de Lyon, Lyon
  - Groupe Hospitalier Region Mulhouse Et Sud Alsace, Mulhouse
  - CHU de Nancy, Nancy
  - Hôpital d'Enfants Armand-Trousseau, Paris
  - Hôpital de la Pitié Salpêtrière, Paris
  - Hôpital Necker Enfants Malades, Paris
  - CHU de Reims, Reims
  - CHU de Rennes, Rennes
  - Les Hôpitaux Universitaires de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided